CLINICAL TRIAL: NCT07153328
Title: Silver Diamine Fluoride in Arresting Dental Caries Among Young Children, a Randomized Clinical Trial
Brief Title: SDF With or Without Fluoride Varnish for Caries Arrest in Primary Teeth of Young Children
Acronym: SDF-FV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaty Dent (Other)
Responsible Party: Principal Investigator, Manola Kelmendi, Principal Investigator; Director- Pediatric Dentistry Unit Beaty Dent Clinic, Beaty Dent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDF-FV-TRIAL-2021-2022; SDF-FV-TRIAL-2021-2022 (Other: Beaty Dent, Tirana, Albania (Sponsor))
Record Dates: First submitted 2025-08-16; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; sodium fluoride topical preparation; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups: (1) semiannual application of 38% silver diamine fluoride (SDF) to active lesions, or (2) an alternating protocol of 38% SDF applied to active lesions and 5% sodium fluoride varnish (FV) applied to all teeth every three months. Participants remained in their assigned group for the 24-month follow-up period.
Who Masked: Outcomes Assessor
Masking Description: No other parties were masked in this study beyond the outcomes assessor, who was blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semiannual 38% Silver Diamine Fluoride (SDF) (Experimental): Participants assigned to this arm receive topical application of 38% silver diamine fluoride (SDF) to all active carious lesions at baseline and every 6 months (months 0, 6, 12, and 18, 24). In addition, a 5% sodium fluoride varnish (NaF) is applied to all teeth at 3-month intervals (months 3, 9, 15, 21). Applications are performed by a dentist using standard microbrush or applicator techniques, ensuring lesions coverage for SDF and full dentition coverage for NaF varnish. This alternating protocol evaluates whether combining periodic SDF with regular fluoride varnish enhances caries arrest in primary teeth compared to semiannual SDF alone.
  Interventions: Drug: Silver Diamine Fluoride (SDF, 38%) and Sodium Fluoride Varnish (NaF, 5%); Drug: Silver Diamine Fluoride (SDF, 38%)
- Alternating 38% SDF + 5% Sodium Fluoride Varnish (FV) (Active Comparator): Participants assigned to this arm receive topical application of 38% silver diamine fluoride (SDF) to all active carious lesions at baseline and every 6 months (months 0, 6, 12, and 18, 24). Applications are performed by a dentist using a microbrush to directly cover the lesion surface until fully saturated. No additional fluoride varnish is provided in this arm. The protocol evaluates the effectiveness of semiannual SDF application alone for arresting active caries in primary teeth of young, uncooperative pediatric patients.
  Interventions: Drug: Silver Diamine Fluoride (SDF, 38%) and Sodium Fluoride Varnish (NaF, 5%)

INTERVENTIONS:
Drug: Silver Diamine Fluoride (SDF, 38%) and Sodium Fluoride Varnish (NaF, 5%) — Application of 38% silver diamine fluoride (SDF) to all active carious lesions at baseline and every 6 months (months 0, 6, 12, and 18, 24). In addition, a 5% sodium fluoride varnish (NaF) is applied to all teeth at 3-month intervals (months 3, 9, 15, 21). Applications are performed by a dentist using standard microbrush or applicator techniques, ensuring lesions coverage for SDF and full dentition coverage for NaF varnish. This alternating protocol evaluates whether combining periodic SDF with regular fluoride varnish enhances caries arrest in primary teeth compared to semiannual SDF alone.
  Other Names: Saforide (Toyo Seiyaku Kasei, Japan), Advantage Arrest (Elevate Oral Care, USA), Riva Star (SDI, Australia), 3M™ Fast Release Varnish, Duraphat (Colgate), CavityShield (3M), Flor-Opal (Ultradent)
Drug: Silver Diamine Fluoride (SDF, 38%) — Application of 38% silver diamine fluoride (SDF) to all active carious lesions at baseline and every 6 months (months 0, 6, 12, and 18, 24). Applications are performed by a dentist using a microbrush to directly cover the lesion surface until fully saturated. No additional fluoride varnish is provided in this arm. The protocol evaluates the effectiveness of semiannual SDF application alone for arresting active caries in primary teeth of young, uncooperative pediatric patients.
  Other Names: Saforide (Toyo Seiyaku Kasei Co., Japan), Advantage Arrest (Elevate Oral Care, USA), Riva Star (SDI Limited, Australia) 3M™ Fast Release Varnish, Duraphat (Colgate-Palmolive), CavityShield
  Arms: Semiannual 38% Silver Diamine Fluoride (SDF)

SUMMARY:
Tooth decay (dental caries) occurs when acids dissolve tooth structure. If not treated, cavities in primary teeth can progress quickly, leading to caries, infection and early tooth loss. These problems may affect chewing, speech, nutrition, and overall health. In Albania and many other countries, cavities in young children are very common. Standard dental treatments are often difficult in very young or uncooperative children and may require sedation or general anesthesia.

Silver diamine fluoride (SDF) is a liquid medication that can be painted directly onto cavities. SDF stops cavities from worsening by killing bacteria and hardening softened tooth surfaces. The main side effect is dark staining of the treated area. Despite this, SDF is considered safe and effective, especially for children who cannot tolerate conventional treatment. Fluoride varnish (FV) is another preventive treatment applied to all tooth surfaces to strengthen enamel and help prevent new cavities.

The purpose of this study is to compare two approaches for managing tooth decay in young children who have difficulty cooperating for dental care:

* SDF applied to cavities every six months.
* SDF applied every six months, with FV applied to all teeth every three months. A total of 104 children between the ages of 1.5 and 8 years with active cavities in their primary (baby) teeth were enrolled. Children were randomly assigned to one of the two treatment groups.

The children were followed for 24 months. The main outcome measured is whether cavities became arrested, meaning the surface became hard and inactive with no further breakdown. Additional outcomes include whether combining SDF with FV provides added benefit and whether baseline factors such as oral hygiene and diet influence treatment success.

The information from this study may help dentists and parents understand how SDF, with or without FV, can be used as a safe, effective, and child-friendly option to manage cavities in young children.

DETAILED DESCRIPTION:
Dental caries is a biofilm-mediated disease driven by dietary sugars and bacterial acid production. The prevalence in primary dentition is high worldwide, especially in low- and middle-income countries. Conventional restorative treatments are difficult to perform in very young or behaviorally uncooperative children, and may require sedation or general anesthesia. Therefore, minimally invasive methods such as silver diamine fluoride (SDF) have gained importance as a practical option for arresting active caries lesions.

Rationale and Objectives SDF (38%) is a topical solution with antimicrobial and remineralizing properties that has been shown to arrest dentin caries in children. A limitation is that it stains carious surfaces black. Fluoride varnish (5% NaF) is widely used as a preventive agent to reduce new caries formation. Combining the two may offer dual benefits: SDF for arresting existing lesions and varnish for preventing new ones. The objective of this randomized clinical trial was to compare the effectiveness of two protocols-SDF alone versus alternating SDF and fluoride varnish-for arresting dentin caries in uncooperative young children with primary teeth.

Study Design This was a two-arm, parallel-group, randomized controlled clinical trial conducted in a pediatric dental setting. A total of 104 children aged 1.5-8 years with at least one active dentin caries lesion in primary teeth were enrolled and randomized in a 1:1 ratio. Children with systemic conditions contraindicating participation were excluded. Informed consent was obtained from parents or guardians, and the protocol was approved by the national ethics committee.

Interventions

Group 1 (SDF only): Lesions received 38% SDF application every 6 months.

Group 2 (SDF + FV): Lesions received 38% SDF application every 6 months, with 5% NaF varnish applied to all teeth every 3 months.

All treatments were delivered by calibrated operators according to standardized protocols. Oral hygiene and dietary advice were given to caregivers.

Outcome Measures

Primary outcome: Caries arrest at 24 months, defined as hardening of the lesion surface with no further progression, assessed visually and tactually by blinded examiners.

Secondary outcomes:

Comparative efficacy between the two protocols

Incidence of new caries in non-treated teeth

Influence of baseline factors (oral hygiene, sugar intake, socioeconomic status) on treatment outcomes

Adverse effects, including pulp symptoms and parental acceptance of staining

Follow-up and Data Collection Clinical examinations were performed at baseline, 6, 12, 18, and 24 months. Standardized diagnostic criteria were used. Lesion depth and activity were recorded, and intra-examiner reliability was periodically tested. Caregivers were interviewed about oral health behaviors. Data were entered into an electronic database with quality control checks.

Statistical Analysis Descriptive statistics were used to summarize baseline characteristics. Caries arrest rates were compared between groups using mixed-effects logistic regression to account for clustering of multiple surfaces within each child. Effect modification by baseline covariates (oral hygiene, sugar intake, socioeconomic status, lesion depth) was tested through interaction terms. Statistical significance was set at p < 0.05. Analyses were performed using Stata software.

Safety and Monitoring SDF and fluoride varnish are approved topical agents for dental use and have well-established safety profiles. Adverse events were monitored and reported. No independent Data Monitoring Committee was appointed given the minimal risk nature of the interventions.

Expected Impact This trial provides comparative evidence on two practical, non-invasive caries management protocols in uncooperative pediatric patients. The findings may inform public health strategies and clinical guidelines for the management of early childhood caries in similar populations.

ELIGIBILITY:
Inclusion Criteria:

Children aged 1.5 to 8 years

Uncooperative to dental procedures (Frankl Behavior Rating 1 or 2)

Presence of at least one active, cavitated carious lesion in primary teeth, without pulp involvement

Eligible primary teeth: active caries without pulp involvement

Exclusion Criteria:

Children with clinical signs of infection (pain, parulis, fistula, or abscess)

Cooperative to dental procedures

Children who are candidates for conscious sedation

Known allergy to silver, fluoride, or ammonia

Teeth with pulpal complications, non-restorable, exfoliating, or scheduled for extraction

Ages: 18 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Caries arrest rate of treated lesions | Baseline, 6, 12, 18, and 24 months post-treatment
  Proportion of active carious lesions that transition to a hardened, non-progressive state (surface hardness on probing, dark discoloration, no cavitation/enlargement), assessed by visual-tactile examination using ICDAS-based criteria under proper lighting and dry conditions. Evaluations conducted by blinded assessors.

SECONDARY OUTCOMES:
Progression of treated lesions to advanced caries or pulpal complications | 6, 12, 18, and 24 months post-treatment
  Proportion of treated surfaces exhibiting progression defined as softened dentin upon probing or development of pulpal complications (pain, parulis/fistula, tenderness to percussion). Lesions meeting failure criteria are withdrawn from arrest analysis and managed according to standard protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Manola Kelmendi, DMD, PhD, Principal Investigator — Faculty of Dental Medicine, University of Medicine of Tirana, Albania; Shirli Kelmendi, PhD Cand., Study Chair — Universidad Cardenal Herrera, UCHCEU, Valencia, Spain
Locations (2):
- Albania (2):
  - Beaty Dent, Tirana, Tirana
  - Happy Dent, Tirana, Tirana

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves pediatric patients, where data protection and confidentiality are paramount. Only aggregate results will be reported in publications.

REFERENCES:
- [Background] Duangthip D, Wong MCM, Chu CH, Lo ECM. Caries arrest by topical fluorides in preschool children: 30-month results. J Dent. 2018 Mar;70:74-79. doi: 10.1016/j.jdent.2017.12.013. Epub 2017 Dec 28. PMID 29289726
- [Background] Trieu A, Mohamed A, Lynch E. Silver diamine fluoride versus sodium fluoride for arresting dentine caries in children: a systematic review and meta-analysis. Sci Rep. 2019 Feb 14;9(1):2115. doi: 10.1038/s41598-019-38569-9. PMID 30765785
- [Background] Abdellatif EB, El Kashlan MK, El Tantawi M. Silver diamine fluoride with sodium fluoride varnish versus silver diamine fluoride in arresting early childhood caries: a 6-months follow up of a randomized field trial. BMC Oral Health. 2023 Nov 17;23(1):875. doi: 10.1186/s12903-023-03597-5. PMID 37978488
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092